CLINICAL TRIAL: NCT03247686
Title: A Phase 2, Double-blind, Placebo-controlled Study of RSLV-132 in Subjects With Primary Sjogren's Syndrome
Brief Title: A Study of RSLV-132 in Subjects With Primary Sjogren's Syndrome
Acronym: RSLV-132
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Resolve Therapeutics (Industry)
Collaborators: University Hospital Birmingham (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 132-04
Record Dates: First submitted 2017-08-03; First posted 2017-08-14 (Actual); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2020-10

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — RSLV-132

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- RSLV-132 (Active Comparator): Experimental drug
  Interventions: Drug: RSLV-132

INTERVENTIONS:
Drug: RSLV-132 — RNase Fc fusion protein
  Arms: RSLV-132
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The present study will examine the role of circulating RNA complexed with autoantibodies and immune complexes and its role in activation of inflammatory pathways in patients with primary Sjogren's syndrome. The study will be conducted in a subset of Sjogren's patients who have elevated levels of autoantibodies and a pattern of elevated interferon-stimulated gene expression in blood cells. A number of biochemical and clinical parameters will be analyzed to determine the potential therapeutic utility of nuclease therapy in Sjogren's syndrome.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, placebo-controlled study to evaluate the impact of 8 intravenous infusions of RSLV-132 in 28 patients with primary Sjogren's syndrome. Each of the subjects will be randomized 3:1 (active:placebo) and will receive 8 infusions of 10 mg/kg of RSLV-132 or placebo as follows on days:

• 1, 8, 15, 29, 43, 57, 71, and 85

Potential subjects will be screened to assess their eligibility to enter the study within 60 days prior to study entry (i.e., prior to Baseline visit). Following Baseline evaluations on Day 1, subjects will receive their first infusion of RSLV-132 or placebo. Subjects will return to the research unit for follow-up visits as described in Appendix A.

Dose selection rationale: The dose level was chosen based on safety and tolerability data from Protocol 132-02 (multiple ascending dose study in SLE patients). Additionally, in a 6-month toxicology study in cynomolgus monkeys, 50 mg/kg of RSLV-132 was administered by IV infusion weekly. No dose-limiting toxicity was noted, therefore the No Observed Adverse Effect Level is at least 50 mg/kg, providing at least a 5-fold safety margin for this study.

RSLV-132 shall be prepared for each subject from individual stock vials provided by Sponsor. Details of dilution, dose preparation, and administration instructions will be provided in the Study Drug Reference Guide. The dose for each individual shall be based on the subject's body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Meet 4 of 6 criteria of 2002 American-European Consensus Group (AECG) criteria for Primary Sjogren's Syndrome
2. Presence of anti Ro autoantibodies
3. Presence of interferon signature

Exclusion Criteria:

1. Use fo hydroxychloroquine within 30 days of baseline
2. Use of cyclophosphamide within 180 days of baseline
3. Use of oral corticosteroids greater than 10 mg/day
4. Known IgG4-related disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Posada, Ph.D., Study Director — Resolve Therapeutics
Locations (2):
- United Kingdom (2):
  - University Hospitals Birmingham, Birmingham, Edgbaston
  - Newcastle upon Tyne Hospitals, Newcastle upon Tyne, Gosforth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Posada J, Valadkhan S, Burge D, Davies K, Tarn J, Casement J, Jobling K, Gallagher P, Wilson D, Barone F, Fisher BA, Ng WF. Improvement of Severe Fatigue Following Nuclease Therapy in Patients With Primary Sjogren's Syndrome: A Randomized Clinical Trial. Arthritis Rheumatol. 2021 Jan;73(1):143-150. doi: 10.1002/art.41489. Epub 2020 Nov 22. PMID 32798283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 12 December 2016 and 01 February 2018. Participants were recruited from the Investigator's medical clinics.
Pre-assignment Details: Participants were randomized in a 3:1 ratio to either RSLV-132 or placebo. A total of 22 participants were randomised to RSLV-2 and 8 to placebo. Two participants randomized to RSLV-2 were withdrawn prior to the start of study treatment, one withdrew consent and one was found not to meet the eligibility criteria.
Period: Overall Study
Arm/Group | Placebo | RSLV-132
Started | 8 | 20
Completed | 7 | 18
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: All participants randomized who received at least one dose of study treatment (RSLV-132 or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | RSLV-132 | Total
Number analyzed (Participants) | 8 | 20 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (8.8) | 56.5 (12.9) | 57.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 20 | 28
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 19 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 19 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 20 | 28
EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The ESSDAI is a systemic disease activity index used in clinical studies. It includes 12 domains (i.e, organ systems: cutaneous, respiratory, renal, articular, muscular, peripheral nervous system, central nervous system, hematological, glandular, constitutional, lymphadenopathic, biological) and each domain is divided into 3 or 4 levels of activity (0 - No, 1 - Low, 2 - Moderate, 3 - High). The score from each domain is added to make the total score. The scale total score ranges from 0 to 123. A lower score represents less disease activity.
  Scores on a scale | 5.1 (4.1) | 5.0 (4.6) | 5.1 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Blood Cell Gene Expression
Description: Interferon gene expression (mean log2 fold change from baseline to Day 99). The of expression of three IFN-inducible genes (HERC5, EPSTI1, CMPK2) was measured by qPCR to assess the IFN signature status (the altered pattern of gene expression) of Sjögren's syndrome patients.
Time Frame: Day 1 and Day 99
Measure: Mean (Standard Error); unit: log 2 fold change
Groups:
- RSLV-132 All: Experimental drug
  RSLV-132: RNase Fc fusion protein
  All participants receiving RSLV-132
- RSLV-132 Responders: Experimental drug
  RSLV-132: RNase Fc fusion protein
  Participants receiving RSLV-132 showing a clinically meaningful improvement in two of the three patient reported outcomes
- RSLV-132 Non-responders: Experimental drug
  RSLV-132: RNase Fc fusion protein
  Participants receiving RSLV-132 not showing a clinically meaningful improvement in two of the three patient reported outcomes
Arm/Group | Placebo | RSLV-132 All | RSLV-132 Responders | RSLV-132 Non-responders
Number analyzed (Participants) | 7 | 20 | 13 | 7
log 2 fold change
  Module M1.2 | -0.0291486 (0.1151235) | 0.1330903 (0.09136563) | 0.2509076 (0.1862489) | 0.06726222 (0.06520814)
  Module M3.4 | -0.0301788 (0.1362689) | 0.08489987 (0.08673372) | 0.1576311 (0.1801423) | 0.0409229 (0.08639682)
  Module M5.12 | -0.0572555 (0.09889587) | 0.02757946 (0.1279434) | 0.0378753 (0.1228119) | 0.0227104 (0.1733785)
Statistical Analysis 1: Comparison: Placebo vs RSLV-132 All; Module M1.2 Placebo versus RSLV-132 All; Test type: Superiority; p = 0.0000496, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs RSLV-132 All; Module M3.4 Placebo versus RSLV-132 All; Test type: Superiority; p = 0.0000103, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo vs RSLV-132 All; Module M5.12 Placebo versus RSLV-132 All; Test type: Superiority; p = 0.0004398, t-test, 2 sided
Statistical Analysis 4: Comparison: Placebo vs RSLV-132 Responders; Module 1.2 Placebo versus RSLV-132 Responders; Test type: Superiority; p = 0.0000068, t-test, 2 sided
Statistical Analysis 5: Comparison: Placebo vs RSLV-132 Responders; Module M3.4 Placebo versus RSLV-132 Responders; Test type: Superiority; p = 0.0000002, t-test, 2 sided
Statistical Analysis 6: Comparison: Placebo vs RSLV-132 Responders; Module 5.12 Placebo versus RSLV-132 Responders; Test type: Superiority; p = 0.0000926, t-test, 2 sided
Statistical Analysis 7: Comparison: Placebo vs RSLV-132 Non-responders; Module M1.2 Placebo versus RSLV-132 Non-responders; Test type: Superiority; p = 0.0015450, t-test, 2 sided
Statistical Analysis 8: Comparison: Placebo vs RSLV-132 Non-responders; Module M3.4 Placebo versus RSLV-132 Non-responders; Test type: Superiority; p = 0.0004632, t-test, 2 sided
Statistical Analysis 9: Comparison: Placebo vs RSLV-132 Non-responders; Module M5.12; Test type: Superiority; p = 0.0096960, t-test, 2 sided

2. Secondary Outcome: EULAR ESSDAI Total Score.
Description: Clinical disease activity: Change from Baseline to Day 99 in European League Against Rheumatism Sjögren's Syndrome Disease Activity Index Total Scores (imputed values with last observation carried forward). The scale ranges from 0 to 123. A higher score means more disease activity (worse outcome).
Time Frame: Days 1, 29, 57, 85 and 99
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | RSLV-132
Number analyzed (Participants) | 8 | 20
Scores on a scale | -2.5 (4.3) | 0.0 (3.8)
Statistical Analysis 1: Comparison: Placebo vs RSLV-132; Mean difference in change from baseline (95% CI); Test type: Equivalence — Two sample t-test with Satterthwaite approximation; p = 0.180, t-test, 2 sided; Mean Difference (Final Values) = -2.50, 95% CI 2-sided [-6.34 to 1.34]

ADVERSE EVENTS:
Time Frame: 211 days
Description: Adverse events were collected from the first dose of study treatment until the last telephone contact on Day 211
Arm/Group | Placebo | RSLV-132
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/20
Other Adverse Events (participants affected / at risk) | 8/8 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | RSLV-132 (N=20)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | RSLV-132 (N=20)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 6 (7)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 3 (4)
Gastoenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 5 (8)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (6)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Palindromic rheumatism (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 3 (4)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sensorimotor disorder (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (2) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03247686/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT03247686/SAP_001.pdf